CLINICAL TRIAL: NCT04191512
Title: Head to Head Comparison of Upper Airway Stimulation and Continuous Positive Airway Pressure; a Pilot Study.
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 19C.245
Record Dates: First submitted 2019-11-22; First posted 2019-12-09 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Upper airway stimulation
- Continuous positive airway pressure

SUMMARY:
To date, there has been no head to head comparison of Upper Airway Stimulation (UAS) and Continuous Positive Airway Pressure (CPAP) utilizing a full night polysomnographic evaluation. With this study we aim to evaluate a pilot cohort of patients with OSA treated with CPAP or UAS using the WatchPAT polysomnography system.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 22 years old
* History of moderate to severe OSA (AHI 15-65)
* UAS implantation with postoperative titration and demonstrated successful use of therapy or has demonstrated the ability to tolerate CPAP for greater than 4 hours per night 5 days per week.

Exclusion Criteria:

* none

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients using upper airway stimulation or continuous positive airway pressure
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-01-21 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Difference in polysomnography (PSG) data between UAS and CPAP groups | 2 years
Difference in Epworth Sleepiness Scale questionnaire data between UAS and CPAP groups | 2 years
Difference in Functional Outcomes of Sleep questionnaire data between UAS and CPAP groups | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Department of Otolaryngology, Philadelphia, Pennsylvania, United States